CLINICAL TRIAL: NCT03742973
Title: A Randomized, Double-Blind, Placebo-Controlled, Proof-of-Concept Study Evaluating the Efficacy and Safety of Baricitinib (LY3009104) in Patients With Primary Biliary Cholangitis Who Have an Inadequate Response or Are Intolerant to UDCA
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Primary Biliary Cholangitis Who do Not Respond or Cannot Take UDCA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to enrollment futility.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17039; I4V-MC-JAIV (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-11-14; First posted 2018-11-15 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2019-10

CONDITIONS: Primary Biliary Cholangitis
Keywords: Janus kinase inhibitor; JAK
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Baricitinib Cohort A (Experimental): Participants received 2 milligram (mg) of Baricitinib tablet orally once a day for 12 weeks. Cohort A is not reported due to protection of personal identifiable information based on enrollment futility.
  Interventions: Drug: Baricitinib
- Placebo Cohort A (Placebo Comparator): Participants received placebo orally once a day for 12 weeks. Cohort A is not reported due to protection of personal identifiable information based on enrollment futility.
  Interventions: Drug: Placebo
- Baricitinib Cohort B (Experimental): Participants received 4 mg of Baricitinib orally once a day for 12 weeks. Cohort B was planned, but due to enrollment futility, the strategic decision was made to terminate the study.
  Interventions: Drug: Baricitinib
- Placebo Cohort B (Placebo Comparator): Placebo administered orally. Cohort B was planned, but due enrollment futility, the strategic decision was made to terminate the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: Baricitinib Cohort A; Baricitinib Cohort B
Drug: Placebo — Administered orally.
  Arms: Placebo Cohort A; Placebo Cohort B

SUMMARY:
This study evaluates the safety and efficacy of baricitinib in participants with primary biliary cholangitis (PBC) who do not respond or are unable to take ursodeoxycholic acid (UDCA).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of PBC (consistent with American Association for the Study of Liver Disease (AASLD) and European Association for Study of the Liver (EASL) Practice Guidelines; as demonstrated by the presence of at least 2 of the following 3 diagnostic factors:

  * History of elevated Alkaline Phosphatase (ALP) levels for at least 6 months
  * Positive antimitochondrial antibodies titer
  * Liver biopsy consistent with PBC
* Have ALP ≥1.67 x ULN but ≤6 x Upper Limit Normal (ULN).
* Taking UDCA for at least 52 weeks (stable dose for at least 12 weeks) prior to Week 0, or have previously taken, but are intolerant (in the opinion of the investigator) to UDCA and have not received UDCA for at least 12 weeks prior to Week 0.
* Nonpregnant, nonbreastfeeding female participants of childbearing potential.

Exclusion Criteria:

* History or presence of other concomitant liver diseases including:

  * Hepatitis C virus (HCV) infection
  * Hepatitis B virus (HBV) infection
  * Primary sclerosing cholangitis
  * Alcoholic liver disease
  * Autoimmune liver disease other than PBC, such as overlap hepatitis
  * Nonalcoholic steatohepatitis
  * Gilbert's syndrome
* Presence of clinical complications of PBC or clinically significant hepatic decompensation, including:

  * Liver transplantation, current placement on a liver transplant list or current Model for End Stage Liver Disease (MELD) score ≥15
  * Portal hypertension with complications, including known gastric or esophageal varices, ascites, history of variceal bleeds or related therapeutic or prophylactic interventions (e.g., beta blockers, insertion of variceal bands or transjugular intrahepatic portosystemic shunt), or hepatic encephalopathy
  * Cirrhosis, including history or presence of one or more of the following:

    * spontaneous bacterial peritonitis
    * hepatocellular carcinoma
  * Hepatorenal syndrome (type I or II)
* Have an estimated glomerular filtration rate (eGFR) based on the most recent available serum creatinine of <90 milliliters/minute/1.73 m2.
* Have screening electrocardiogram (ECG) abnormalities that in the opinion of the investigator or the sponsor are clinically significant and indicate an unacceptable risk for the participant's participation in the study.
* Have experienced any of the following within 12 weeks of screening: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of venous thromboembolism (VTE) (deep vein thrombosis/pulmonary embolism [DVT/PE]).
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
* Have a current or recent (<4 weeks prior to randomization) clinically serious infection or any other active or recent infection that, in the opinion of the investigator, would pose an unacceptable risk to the participant if participating in the study.
* Have had symptomatic herpes zoster infection within 12 weeks prior to randomization.
* Have active tuberculosis (TB) disease determined on the basis of a positive medical history, physical examination, or chest radiography (per local standard of care) or latent TB infection (LTBI).
* Have any of the following specific abnormalities based on screening central lab test results:

  * Hemoglobin <10 grams per deciliter (100.0 grams per liter)
  * Alanine aminotransferase (ALT) >3 x ULN
  * aspartate aminotransferase (AST) >3 x ULN
  * alkaline phosphatase (ALP) >6 x ULN
  * Total bilirubin level (TBL) >ULN
  * Creatine phosphokinase (CPK) > ULN
  * Serum albumin < lower limit of normal (LLN)
  * International Normalized Ratio of Prothrombin Time (INR) > ULN
  * Total white blood cell (WBC) count <LLN
  * Absolute neutrophil count (ANC) <LLN
  * Lymphocyte count <LLN
  * Platelet (thrombocyte) count <LLN
* Are receiving unstable treatment for pruritus within 6 weeks prior to Week 0.
* Have been treated with systemic (oral or parenteral) corticosteroids within 6 weeks prior to Week 0.
* Have received biologic treatments for an immunologic disease within 4 weeks of screening.
* Have received a Janus kinase (JAK) inhibitor.
* Have received obeticholic acid.
* Have received fenofibrate or other fibrates for the treatment of PBC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (10):
  - Southern California GI and Liver Centers (SCLC), Coronado, California
  - University of California, Davis - Health Systems, Sacramento, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - The Institute for Digestive Health and Liver Disease at Mercy, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - NYU Langone, New York, New York
  - UH Cleveland Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- Puerto Rico (2):
  - Klinical Investigations Group, LLC, San Juan, PR
  - University of Puerto Rico, Medical Sciences Campus, San Juan, PR

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org

REFERENCES:
- See also: Click here for more information about this study: A Study of Baricitinib (LY3009104) in Participants With Primary Biliary Cholangitis Who do Not Respond or Cannot Take UDCA — https://www.lillytrialguide.com/en-US/studies/liver-disease/JAIV#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Zero participants reported in cohort A due to protection of personal identifiable information based on enrollment futility and cohort B is not reported due to early study termination based on enrollment futility.
Groups:
- Baricitinib Cohort A: Participants received 2 milligram (mg) of Baricitinib tablet orally once a day for 12 weeks.
- Placebo Cohort A: Participants received placebo orally once a day for 12 weeks.
Period: Overall Study
Arm/Group | Baricitinib Cohort A | Placebo Cohort A
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero participants reported in cohort A due to protection of personal identifiable information based on enrollment futility.
Groups:
- .Baricitinib Cohort A: Participants received 2 mg of Baricitinib tablet orally once a day for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort A | .Baricitinib Cohort A | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment
Baseline in ALP [unit: microgram/Liter (u/L)]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alkaline Phosphatase (ALP)
Description: Change from baseline in Alkaline Phosphatase (ALP)
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Groups:
- Baricitinib Cohort A: Participants received 2 mg of Baricitinib tablet orally once a day for 12 weeks.
Arm/Group | Baricitinib Cohort A | Placebo Cohort A
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Alkaline Phosphatase (ALP) <1.67 x Upper Limit of Normal (ULN) (and at Least 15% Decrease From Baseline) and Total Bilirubin Level Less Than ULN
Description: Percentage of participants with alkaline phosphatase (ALP) <1.67 x Upper Limit of Normal (ULN) (and at least 15% decrease from baseline) and total bilirubin level less than ULN.
Time Frame: Week 12
Population: Zero participants with evaluable data was reported in cohort A due to protection of personal identifiable information based on enrollment futility.
Arm/Group | Baricitinib Cohort A
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Itch Numeric Rating Scale (NRS)
Description: Change from baseline in itch NRS. The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by circling the number that best describes the worst level of itching in the past 7 days.
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Arm/Group | Baricitinib Cohort A | Placebo Cohort A
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Fatigue NRS
Description: Change from baseline in fatigue NRS. The Fatigue NRS is a single-item, patient-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine." Overall severity of a participant's fatigue is indicated by selecting the number that describes the worst level of fatigue during the past 7 days.
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Arm/Group | Baricitinib Cohort A | Placebo Cohort A
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 Months
Description: Zero participants reported in cohort A due to protection of personal identifiable information based on enrollment futility and cohort B is not reported due to early study termination based on enrollment futility.
Arm/Group | Baricitinib Cohort A | Placebo Cohort A
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Zero participants reported in cohort A due to protection of personal identifiable information based on enrollment futility and cohort B is not reported due to early study termination based on enrollment futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT03742973/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT03742973/SAP_001.pdf